CLINICAL TRIAL: NCT01996072
Title: A Pilot & Feasibility Study of the Imaging Potential of EC17 in Subjects Undergoing Parathyroidectomy for Primary Hyperparathyroidism.
Brief Title: EC17 for Intraoperative Imaging for Parathyroidectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sunil Singhall, Assistant Proffesor of Medicine, Assistant Proffesor of Surgery, Director Thoracic Surgery Research Lab, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 818060; 818060 [UPenn IRB Protocol] (Other: IRB)
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Primary Hyperparathyroidism
Keywords: Primary hyperparathyroidism; Parathyroid
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EC17 Injection Group (Experimental): The group will receive a single dose of EC17, infused over 10 minutes, prior to surgery. Then, during surgery, the EC-17 will be imaged with a camera that the investigators have developed.
  Interventions: Drug: EC17

INTERVENTIONS:
Drug: EC17
  Other Names: Folate- FITC

SUMMARY:
Primary hyperparathyroidism is a significant medical and public health problem in the world and affects approximately 100,000 new patients in the United States alone. If left untreated this can lead to renal stones, osteoporosis, fatigue, and depression. The best treatment for primary hyperparathyroidism is surgical parathyroidectomy. However surgical parathyroidectomy can be difficult due to the variant location of the parathyroid glands. Up to 5% of patients leave the operating room without surgical cure.

Primary hyperparathyroidism is an ideal disease to investigate intraoperative fluorescent imaging. This would allow surgeons to identify the parathyroid glands and resect the suspicious parathyroid glands. Folate receptor (FR) has been found to be over-expressed in parathyroid tissue and not thyroid issues. An ideal surgical treatment would combine FR-specific fluorescent tracers with intraoperative imaging. It is important to note that FR is expressed only in the proximal tubules of the kidneys, activated macrophages, and in the choroidal plexus. Thus, the false positive detection rate is expected to be extremely low.

A group well known to us in the Netherlands has completed a pilot study utilizing a folate-FITC conjugate in 12 patients with ovarian cancer. Another group of investigators in Mayo have subsequently performed this study on 20 more patients without any serious adverse events (personal communication). They report excellent sensitivity and specificity with this technique with only grade 1 side effects (allergic reaction). All side effects reversed when the injection was halted. Patients with a history of allergic reactions to insect bites should not participate (fluorescein is derived from the firefly insect, folate is an essential vitamin).

A fluorescent contrast agent (folate-FITC or EC17) will be used to determine if it will localize to the primary tumor nodule(s) or mass(es) of patients undergoing parathyroid surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 18 years of age
2. Patients presenting with primary hyperparathyroidism presumed to be resectable on pre-operative assessment
3. Good operative candidate
4. Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria:

1. Pregnant women as determined by urinary or serum beta hCG within 72 hours of surgery
2. Patients with a history of anaphylactic reactions to Folate-FITC or insects
3. Vulnerable patient populations

   1. Homeless patients
   2. Patients with drug or alcohol dependence
   3. Children and neonates
   4. Patients unable to participate in the consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The ability of EC17 and the imaging system to detect FRA positive tumors during surgery conducted 2-4 hours post EC-17 administration. | Within two to four hours of injection of EC17

SECONDARY OUTCOMES:
The number of participants that will have an adverse reaction to EC17 | Day 1-Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States